CLINICAL TRIAL: NCT00874107
Title: A Phase 2, Randomized, Efficacy and Safety Study of Imprime PGG® Injection in Combination With Bevacizumab and Concomitant Paclitaxel and Carboplatin Therapy in Patients With Previously Untreated Advanced (Stage IIIB or IV) Non-Small Cell Lung Cancer
Brief Title: Efficacy/Safety of Imprime PGG® Injection With Bevacizumab and Paclitaxel/Carboplatin in Patients With Untreated Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HiberCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-CL-PGG-LCA0821
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Phase 2; Randomized; Efficacy; Safety; Imprime PGG; Bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Imprime PGG + bevacizumab + paclitaxel/carboplatin
  Interventions: Biological: Imprime PGG® Injection; Biological: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin
- 2 (Other): bevacizumab + paclitaxel/carboplatin
  Interventions: Biological: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: Imprime PGG® Injection — 4 mg/kg, i.v. over 2 hr, weekly until progression or discontinuation
  Arms: 1
Biological: Bevacizumab — 15 mg/kg, i.v., over 90 minutes, on Day 1 only of each 3-week treatment cycle
Drug: Paclitaxel — 200 mg/m2, i.v. over 3 hr, on Day 2 of each 3-week treatment cycle for the first 4 to 6 treatment cycles.
Drug: Carboplatin — AUC of 6 mg./mL · min based on the Calvert formula; i.v. over 30 min, on Day 2 of each 3-week treatment cycle for the first 4 to 6 treatment cycles

SUMMARY:
The Phase 2 study described in this protocol will serve to evaluate the antitumor activity, safety and pharmacokinetic profile of Imprime PGG when combined with bevacizumab and concomitant paclitaxel and carboplatin therapy in patients with previously untreated advanced NSCLC. Additionally, this study will provide guidance for the design of more definitive efficacy studies of Imprime PGG in NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Has read, understood and signed the informed consent form (ICF) approved by the Independent Review Board/Ethics Committee (IRB/EC);
2. Is between the ages of 18 and 75 years old, inclusive;
3. Has histologically or cytologically confirmed stage IIIB (malignant pericardial or pleural effusion) or stage IV non-small cell lung cancer;
4. Has non-squamous, non-small cell lung cancer
5. Has measurable disease, defined as at least one tumor that fulfills the criteria for a target lesion according to RECIST;
6. Has an ECOG performance status of 0 or 1;
7. Has a life expectancy of > 3 months;
8. Has adequate hematologic function as evidenced by:

   1. ANC ≥ 1,500/μL
   2. PLT ≥ 100,000/μL
   3. HGB ≥ 9 g/dL obtained within 1 week prior to the first dose of study medication;
9. Has adequate renal function as evidenced by:

   1. Serum creatinine ≤ 1.5 X the upper limit of normal (ULN) for the reference lab
   2. Urine dipstick for proteinuria of < 1+ (i.e., either 0 or trace) within 2 weeks of Day 1 If urine dipstick is ≥ 1+, then urine protein excretion must be ≤ 500 mg over a 24 hour collection obtained within 1 week prior to the first dose of study medication;
10. Has adequate hepatic function as evidenced by:

    1. Serum total bilirubin ≤ 1.0 mg/dL
    2. AST ≤ 2.5X ULN for the reference lab (≤ 5X ULN for subjects with known hepatic metastases)
    3. ALT ≤ 2.5X ULN for the reference lab (≤ 5X ULN for subjects with known hepatic metastases) obtained within 1 week prior to the first dose of study medication;
11. Has adequate coagulation function as evidenced by:

    1. INR ≤ 1.5
    2. PTT ≤ ULN for the reference lab obtained within 1 week prior to the first dose of study medication;
12. If a woman of childbearing potential or a fertile man (and his partners), must agree to use an effective form of contraception (hormonal contraceptive, double-barrier method or abstinence) during the study.

Exclusion Criteria:

1. Has received prior systemic chemotherapy at any time for lung cancer;
2. Has received previous radiation therapy to >30% of active bone marrow or any radiation therapy within 3 weeks of Day 1;
3. Has a known hypersensitivity to baker's yeast, or has an active yeast infection;
4. Has had previous exposure to Betafectin® or Imprime PGG;
5. Has an active infection;
6. Presents with any of the following medical diagnoses/conditions at the time of screening:

   1. Central nervous system (CNS) metastases
   2. Uncontrolled hypertension (>150/100 mmHg) or hypertension that requires > two agents for adequate control
   3. Peripheral neuropathy ≥ grade 2 from any cause
   4. Fever of >38.5° C within 3 days prior to screening or Day 1, initial dosing
   5. Known HIV/AIDs, Hepatitis B, Hepatitis C, connective tissue or autoimmune disease, or other clinical diagnosis, ongoing or intercurrent illness that in the physician's opinion could interfere with participation
7. Has a history of any of the following medical diagnoses/conditions:

   1. Arterial or venous thromboembolic or hemorrhagic disorders including stroke, transient ischemic attack or cerebral infarction
   2. Deep vein thrombosis within 1 year prior to screening
   3. Myocardial infarction or an unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure) within the previous 6 months
   4. Second malignancy within the previous 5 years, other than basal cell carcinoma, cervical intra-epithelial neoplasia or curatively treated prostate cancer with a PSA of <2.0 ng/mL
8. Has a known hypersensitivity to bevacizumab, murine proteins, or any component of bevacizumab;
9. Has a know sensitivity to polyethoxylated castor oil;
10. Has previously received treatment with bevacizumab;
11. Has had surgery within 4 weeks of Day 1 or needle or open biopsy within 1 week of Day 1;
12. Has a non-healing wound or gastric ulcer;
13. Has a non-healed bone fracture;
14. Is receiving systemic anti-coagulation therapy (e.g., dipyridalmole (Persantine®), ticlopidine (Ticlid®), clopidogrel (Plavix®) and /or cilostazol (Pletal®);
15. Is receiving chronic daily treatment with aspirin (>100 mg/day) or other nonsteroidal anti-inflammatory agents known to inhibit platelet function within 1 week of Day 1;
16. Presents with any of the following medical diagnoses/conditions at the time of screening:

    a. Predominant squamous cell histology
17. Has a history of any of the following medical diagnoses/conditions:

    1. Hemoptysis (≥ ½ tsp red blood)
    2. Bleeding diathesis or coagulopathy
18. If female, is pregnant or breast-feeding;
19. Is receiving concurrent investigational therapy or has received investigational therapy within a period of 30 days prior to the first scheduled day of dosing (investigational therapy is defined as treatment for which there is currently no regulatory-authority-approved indication);
20. Has previously received an organ or progenitor/stem cell transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-06; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To determine the objective response rate (ORR) in each study arm | Approximately 1.5 years

SECONDARY OUTCOMES:
To determine the disease control rate (DCR) in each study arm | Approximately 1.5 years
To determine the complete response (CR), partial response (PR), and stable disease (SD) rates in each study arm | Approximately 1.5 years
To determine the duration of objective tumor response in each study arm | Approximately 1.5 years
To determine the duration of stable disease in each study arm | Approximately 1.5 years
To determine the duration of time to progression (TTP) in each study arm | Approximately 1.5 years
To assess the safety of the dosing regimen within each study arm | Approximately 1.5 years
To determine the pharmacokinetic (PK) profile of Imprime PGG (in active treatment arm only) | Approximately 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Folker Schneller, MD, Principal Investigator — Klinikum rechts der Isar der Technischen Universitaet Muenchen
Locations (10):
- United States (3):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Gabrail Cancer Center, Canton, Ohio
  - University of Texas Health Science Center, San Antonio, San Antonio, Texas
- Germany (7):
  - Kliniken der Stadt Köln gGmbH, Cologne
  - Hospital Marth-Maria Halle Dolau, Halle
  - Clinical Kassel GmbH, Kassel
  - University of Mainz, Mainz
  - University of Munich, Munich
  - Pius-Hospital Oldenburg, Oldenburg
  - Universitätsklinikum Ulm, Ulm

REFERENCES:
- [Background] Salvador C, Li B, Hansen R, Cramer DE, Kong M, Yan J. Yeast-derived beta-glucan augments the therapeutic efficacy mediated by anti-vascular endothelial growth factor monoclonal antibody in human carcinoma xenograft models. Clin Cancer Res. 2008 Feb 15;14(4):1239-47. doi: 10.1158/1078-0432.CCR-07-1669. PMID 18281559
- [Derived] Engel-Riedel W, Lowe J, Mattson P, Richard Trout J, Huhn RD, Gargano M, Patchen ML, Walsh R, Trinh MM, Dupuis M, Schneller F. A randomized, controlled trial evaluating the efficacy and safety of BTH1677 in combination with bevacizumab, carboplatin, and paclitaxel in first-line treatment of advanced non-small cell lung cancer. J Immunother Cancer. 2018 Feb 27;6(1):16. doi: 10.1186/s40425-018-0324-z. PMID 29486797